CLINICAL TRIAL: NCT00456937
Title: Escitalopram in the Treatment of Patient Suffering From Scizophrenia and Obsessive Compulsive Disorder- an Open Label Study
Brief Title: Escitalopram in Schizophrenia in OCD- Open Label Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: BeerYaakov Mental Health Center (Other Government)
Collaborators: Lundbeck Israel (Industry)
Responsible Party: Dr Rafael Stryjer, Beer-Yaakov MHC
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: Escitalopram-173CTIL
Record Dates: First submitted 2006-12-03; First posted 2007-04-05 (Estimated); Last update posted 2009-01-27 (Estimated); Status verified 2009-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Escitalopram

SUMMARY:
SSRI's has been demonstrated to be partially effective in schizophrenia and OCD. We therefore suggest that Escitalopram up to 20 mg /d in those patients could be effective in reducing obsessive compulsive symptomatology

ELIGIBILITY:
Inclusion Criteria:

* Patients who suffer from schizophrenia and OCD

Exclusion Criteria:

* Substance abuse,
* Serious medical condintions,
* Being on SSRI treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Octavio Stryjer, M.D., Principal Investigator — Beer Yaakov Mental Health Center
Locations (1):
- Beer Yaakov MHC, Beer Yaakov, Israel